CLINICAL TRIAL: NCT06769620
Title: A Phase 1, Randomized, Double-blind, Placebo-Controlled, Single-Ascending-Dose Study to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of Intravenous ORT247 in Healthy Volunteers
Brief Title: A First in Human Study of ORT247 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orthogonal Neuroscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ORT247-001
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: After screening, eligible subjects will be enrolled into 1 of 5 planned cohorts: 75 mg, 150 mg, 300 mg, 600 mg, and 1200 mg. The study will start with the lowest dose cohort, and each dose cohort will consist of 8 subjects (6 active, 2 placebo). A safety review committee consisting of the sponsor's medical director, the contract research organization's (CRO's) medical monitor, and the site principal investigator will review AE data collected after dosing to evaluate the following:
  1. Acceptability of proceeding with enrollment of the full cohort of 8 subjects based on review of safety data of the initial 2 subjects (sentinels: 1 active, 1 placebo) through 48 hours after dosing
  2. Acceptability of proceeding with enrollment of the subsequent cohort and studying ascending doses based on review of data for the full cohort of 8 subjects (6 active, 2 placebo) through 7 days after dosing and ongoing data from prior cohorts.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ORT247 (Experimental): Single ascending dose of intravenous ORT247 administered as a infusion over 60 minutes. Subjects enrolled into 1 of 5 planned cohorts will receive 75mg, 150mg, 300mg, 600mg, and 1200mg with dosing being conducted in a staggered fashion, separated by at least 30 minutes of an infusion in one subject and the start of an infusion in another subject.
  Interventions: Drug: ORT247
- Placebo (Placebo Comparator): Single intravenous dose of vehicle with dosing being conducted in a staggered fashion, separated by at least 30 minutes of an infusion in one subject and the start of an infusion in another subject.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORT247 — ORT247 will be provided to study sites in single-use, sterile vials for infusion. Each dose will be prepared with normal saline for infusion.
  Arms: ORT247
Drug: Placebo — Placebo consists of normal saline
  Arms: Placebo

SUMMARY:
This is a single center, double-blinded, randomized, placebo controlled single ascending dose clinical study, with the primary purpose of evaluating the safety, tolerability, pharmacokinetics (PK), and immunohistochemistry of escalating intravenous doses of ORT247 in healthy volunteers.

DETAILED DESCRIPTION:
This is a phase 1, first in human, study of ORT247

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily consents to participate in this study and provides written informed consent before the start of any study-specific procedures
* Male and females, 18 to 65 years of age at time of screening

  1. Female subjects of childbearing potential must not be breastfeeding and must have no plans to become pregnant during the course of the study through 120 days after infusion of study drug. Female subjects of childbearing potential who are heterosexual must agree to use a method of contraception considered to be highly effective (i.e., results in <1% failure rate when used consistently and correctly) from screening through 120 days after the last dose of study drug
  2. Female subjects of non-childbearing potential must have evidence from their medical history indicating that they are not of childbearing potential and must not currently be breastfeeding.
* Any non-vasectomized male subjects must have agreed to use barrier contraceptives plus spermicide for 200 days after dosing.
* Male subjects must agree not to donate sperm for 200 days after dosing
* Female subjects must agree not to preserve eggs (ova) for 120 days after dosing
* Has not participated in a clinical drug study within 30 days of study start, or within 5 half-lives, unless study blind has been broken and the subject was known to be on placebo
* Body mass index of 18-32

Exclusion Criteria:

* Contraindication to undergo LP including international normalized ratio (INR) >1.4 or other coagulopathy, platelet cell count of <120,000/μL, infection at the desired LP site, current use of anti-coagulant medication except for low dose aspirin, degenerative arthritis, spinal scoliosis, back surgery, suspected increased intracranial pressure on history or neurologic exam, non-communicating hydrocephalus or intracranial mass, or prior history of spinal mass or trauma
* Any significant acute or chronic medical illness
* Any history of cancer within 5 years of enrollment with the exception of resected skin basal cell carcinoma
* Any major surgery within 4 weeks of study drug administration
* Donation of blood or serum >500 mL to a blood bank or in a clinical study (except screening visit) within 3 months of study drug administration
* Inability to undergo venipuncture or tolerate venous access
* Has smoked or used tobacco products within 3 months before study drug administration
* Positive drug screen for alcohol, drugs of abuse, or tobacco
* Recent (within 6 months of study drug administration) drug or alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V), Diagnostic Criteria for Drug and Alcohol Abuse
* Evidence of any clinically significant neurological or psychiatric disorder that could interfere with study assessments as determined by investigator and sponsor
* History of or currently has schizophrenia, schizoaffective disorder or bipolar disorder, untreated major depression (DSM-V or International Statistical Classification of Diseases and Related Health Problems, 10th edition [ICD-10] criteria)
* Significant illness or infection requiring intervention within the prior 30 days as determined by investigator and sponsor (must test negative for active coronavirus disease 2019 [COVID-19])
* Indication of potential suicidality risk
* Any of the following abnormalities at screening: serum creatinine > upper limit of normal (ULN), hepatic transaminases (aspartate aminotransferase or alanine aminotransferase) > ULN, abnormal blood pressure based on the clinical judgment of the investigator, QTcF >470 msec
* Known history of hypersensitivity to any component of the ORT247 drug product or placebo
* Currently taking, or planning to take, any medication (prescription or over-the-counter) that would potentially affect the assessment of pharmacokinetics (PK), pharmacodynamics (PD), or immunogenicity of ORT247.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events assessed by severity, frequency and causality | From enrollment to day 85 or early termination

SECONDARY OUTCOMES:
Time to maximum observed serum concentration (Tmax) | Before and at end of infusion (0 hours), and 0.5, 1, 2, 4, 8, and 12, 24, 36 and 48 hours after infusion. Additional samples for assessment of serum concentrations were collected on Day 8, 15, 29, 43, 57, 71 and 85/early termination.
Maximum observed serum concentration (Cmax) | Before and at end of infusion (0 hours), and 0.5, 1, 2, 4, 8, and 12, 24, 36 and 48 hours after infusion. Additional samples for assessment of serum concentrations were collected on Day 8, 15, 29, 43, 57, 71 and 85/early termination.
Number of subjects developing anti-drug antibodies | From enrollment to day 85 or early termination
  Titer and neutralizing activity of anti-drug antibodies will be evaluated
Area under the curve from Time 0 to 168 hours (AUC0-168) | Before and at end of infusion (0 hours), and 0.5, 1, 2, 4, 8, and 12, 24, 36 and 48 hours after infusion. Additional samples for assessment of serum concentrations were collected on Day 8, 15, 29, 43, 57, 71 and 85/early termination.
Area under the curve from Time 0 to last sampling time (AUC0-t) | Before and at end of infusion (0 hours), and 0.5, 1, 2, 4, 8, and 12, 24, 36 and 48 hours after infusion. Additional samples for assessment of serum concentrations were collected on Day 8, 15, 29, 43, 57, 71 and 85/early termination.
Area under the curve from Time 0 to infinity (AUC0-∞) | Before and at end of infusion (0 hours), and 0.5, 1, 2, 4, 8, and 12, 24, 36 and 48 hours after infusion. Additional samples for assessment of serum concentrations were collected on Day 8, 15, 29, 43, 57, 71 and 85/early termination.
Time to clearance (CL) following single i.v. infusion of ORT247 | Before and at end of infusion (0 hours), and 0.5, 1, 2, 4, 8, and 12, 24, 36 and 48 hours after infusion. Additional samples for assessment of serum concentrations were collected on Day 8, 15, 29, 43, 57, 71 and 85/early termination.
Volume of distribution (Vd) following single i.v. infusion of ORT247 | Before and at end of infusion (0 hours), and 0.5, 1, 2, 4, 8, and 12, 24, 36 and 48 hours after infusion. Additional samples for assessment of serum concentrations were collected on Day 8, 15, 29, 43, 57, 71 and 85/early termination.
Terminal half-life (t1/2) following single i.v. infusion of ORT247 | Before and at end of infusion (0 hours), and 0.5, 1, 2, 4, 8, and 12, 24, 36 and 48 hours after infusion. Additional samples for assessment of serum concentrations were collected on Day 8, 15, 29, 43, 57, 71 and 85/early termination.

OTHER OUTCOMES:
Cerebrospinal Fluid Concentrations of ORT247 following single i.v. infusion | Day 3
Concentrations of ORT247 in skeletal muscle biopsy tissue | Day 2
Localization of ORT247 at neuromuscular junctions from skeletal muscle biopsies using immunohistochemistry | Day 2
Ratio of pEphA4 to total EphA4 in human peripheral blood mononuclear cells (PMBC) and skeletal muscle biopsies as a measure of pharmacodynamic activity | PMBC: Baseline, Day 2, and Day 29. Skeletal Muscle Biopsy: Day 2
  Ephrin Type-A Receptor 4 (EphA4) is protein coding gene that interacts with Ephrin ligands and regulates various biological processes in the nervous system

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No